CLINICAL TRIAL: NCT06508164
Title: International Calcium Release Deficiency Syndrome Registry
Brief Title: International CRDS Registry
Acronym: CRDS Registry
Status: Recruiting | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16861
Record Dates: First submitted 2024-07-08; First posted 2024-07-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Calcium Release Deficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 26 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CRDS: Possesses a rare RYR2 variant characterized to be loss-of-function based on in vitro testing consistent with a CRDS diagnosis
- Carrier of an RYR2 truncating variant or large copy number variant: Possesses a rare RYR2 truncating variant and/or large copy number variant involving the RYR2 gene.
- Carrier of a non-functional RYR2 rare variant: Possesses a rare RYR2 variant that is NOT loss-of-function based on in vitro testing and has a clinical phenotype that was considered compatible with CRDS

SUMMARY:
Calcium Release Deficiency Syndrome (CRDS) is a newly discovered genetic arrhythmia syndrome that confers a risk of life-threatening arrhythmias secondary to RYR2 loss-of-function. The International CRDS registry has been designed to facilitate large-scale evaluation of CRDS, including its phenotypic spectrum, approaches to risk stratification, and optimal treatment strategies.

DETAILED DESCRIPTION:
Calcium Release Deficiency Syndrome (CRDS) is a recently discovered inherited arrhythmia syndrome that predisposes to malignant ventricular arrhythmias and sudden cardiac death (SCD). The underlying genetic culprit of CRDS is RYR2, which encodes the cardiac ryanodine receptor. In contrast to Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT), which stems from pathogenic RYR2 gain-of-function, CRDS manifests secondary to RyR2 loss-of-function. Enrolment into the CRDS registry requires that the putative disease causing RYR2 variant is confirmed to result in a loss-of-function on in vitro functional analysis. Individuals possessing an RYR2 truncating variant or large copy number variant will be eligible for enrolment into a second registry arm. Patients with a suspected CRDS diagnosis whose RYR2 variant is found not to impact function will be entered into a control arm of the registry.

Given its recent discovery, our understanding of CRDS remains in its infancy. The International CRDS registry has been designed to facilitate evaluation of large numbers of CRDS patients and enable robust insights to hopefully improve management of affected patients and families.

ELIGIBILITY:
CRDS Cohort

Inclusion Criterion:

- Presence of a rare* RYR2 variant that is characterized to be loss-of-function based on in vitro testing#

RYR2 Truncating and Large CNV Cohort

Inclusion Criterion:

- Presence of a rare* RYR2 truncating variant and/or large copy number variant involving the RYR2 gene.

Carriers of a Non-Functional RYR2 variant

Inclusion Criterion:

- Presence of a rare* RYR2 variant that is characterized to be neither loss- nor gain-of-function based on in vitro testing#

*rare defined as gnomAD prevalence < 0.1%

#RYR2 in vitro functional testing will be performed in the laboratory of Dr. Wayne Chen (University of Calgary)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry will enrol 3 separate cohorts. The primary cohort consists of CRDS cases. A CRDS case is defined as an individual that possesses a rare RYR2 variant proven to be loss-of-function on in vitro analysis. A second cohort consists of individuals that possess a rare RYR2 truncating variant or large copy number variant. The third cohort involves individuals suspected of having CRDS, however in vitro analysis revealed that their rare RYR2 variant did not impact function.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Malignant Ventricular Arrhythmia | 5 years
  Composite of malignant syncope, ICD shock, cardiac arrest, and sudden cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Roston, MD, PhD, Study Chair — University of British Columbia; Jason D Roberts, MD MAS, Principal Investigator — McMaster University; SR Wayne Chen, PhD, Principal Investigator — University of Calgary
Locations (16):
- United States (3):
  - University of California, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
- Garvan Institute of Medical Research, Darlinghurst, New South Wales, Australia
- Belgium (2):
  - Antwerp University Hospital, Edegem, Antwerp
  - Universitair Ziekenhuis Brussel, Brussels
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Montréal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec-Université Laval, Québec, Quebec
- Aarhus University Hospital, Aarhus, Denmark
- CHU de Bordeaux, Bordeaux, Nouvelle-Aquitaine, France
- Shaare Zedek Medical Center, Jerusalem, Israel
- City St George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun B, Yao J, Ni M, Wei J, Zhong X, Guo W, Zhang L, Wang R, Belke D, Chen YX, Lieve KVV, Broendberg AK, Roston TM, Blankoff I, Kammeraad JA, von Alvensleben JC, Lazarte J, Vallmitjana A, Bohne LJ, Rose RA, Benitez R, Hove-Madsen L, Napolitano C, Hegele RA, Fill M, Sanatani S, Wilde AAM, Roberts JD, Priori SG, Jensen HK, Chen SRW. Cardiac ryanodine receptor calcium release deficiency syndrome. Sci Transl Med. 2021 Feb 3;13(579):eaba7287. doi: 10.1126/scitranslmed.aba7287. PMID 33536282
- [Background] Roston TM, Wei J, Guo W, Li Y, Zhong X, Wang R, Estillore JP, Peltenburg PJ, Noguer FRI, Till J, Eckhardt LL, Orland KM, Hamilton R, LaPage MJ, Krahn AD, Tadros R, Vinocur JM, Kallas D, Franciosi S, Roberts JD, Wilde AAM, Jensen HK, Sanatani S, Chen SRW. Clinical and Functional Characterization of Ryanodine Receptor 2 Variants Implicated in Calcium-Release Deficiency Syndrome. JAMA Cardiol. 2022 Jan 1;7(1):84-92. doi: 10.1001/jamacardio.2021.4458. PMID 34730774
- [Background] Li Y, Wei J, Guo W, Sun B, Estillore JP, Wang R, Yoruk A, Roston TM, Sanatani S, Wilde AAM, Gollob MH, Roberts JD, Tseng ZH, Jensen HK, Chen SRW. Human RyR2 (Ryanodine Receptor 2) Loss-of-Function Mutations: Clinical Phenotypes and In Vitro Characterization. Circ Arrhythm Electrophysiol. 2021 Sep;14(9):e010013. doi: 10.1161/CIRCEP.121.010013. Epub 2021 Sep 1. PMID 34546788
- [Background] Ormerod JOM, Ormondroyd E, Li Y, Taylor J, Wei J, Guo W, Wang R, Sarton CNS, McGuire K, Dreau HMP, Taylor JC, Ginks MR, Rajappan K, Chen SRW, Watkins H. Provocation Testing and Therapeutic Response in a Newly Described Channelopathy: RyR2 Calcium Release Deficiency Syndrome. Circ Genom Precis Med. 2022 Feb;15(1):e003589. doi: 10.1161/CIRCGEN.121.003589. Epub 2021 Dec 24. PMID 34949103
- [Background] Ni M, Li Y, Wei J, Song Z, Wang H, Yao J, Chen YX, Belke D, Estillore JP, Wang R, Vallmitjana A, Benitez R, Hove-Madsen L, Feng W, Chen J, Roston TM, Sanatani S, Lehman A, Chen SRW. Increased Ca2+ Transient Underlies RyR2-Related Left Ventricular Noncompaction. Circ Res. 2023 Jul 7;133(2):177-192. doi: 10.1161/CIRCRESAHA.123.322504. Epub 2023 Jun 16. PMID 37325910
- [Background] Ni M, Dadon Z, Ormerod JOM, Saenen J, Hoeksema WF, Antiperovitch P, Tadros R, Christiansen MK, Steinberg C, Arnaud M, Tian S, Sun B, Estillore JP, Wang R, Khan HR, Roston TM, Mazzanti A, Giudicessi JR, Siontis KC, Alak A, Acosta JG, Divakara Menon SM, Tan NS, van der Werf C, Nazer B, Vivekanantham H, Pandya T, Cunningham J, Gula LJ, Wong JA, Amit G, Scheinman MM, Krahn AD, Ackerman MJ, Priori SG, Gollob MH, Healey JS, Sacher F, Nof E, Glikson M, Wilde AAM, Watkins H, Jensen HK, Postema PG, Belhassen B, Chen SRW, Roberts JD. A Clinical Diagnostic Test for Calcium Release Deficiency Syndrome. JAMA. 2024 Jul 16;332(3):204-213. doi: 10.1001/jama.2024.8599. PMID 38900490